CLINICAL TRIAL: NCT01713712
Title: Ease of Access to Nutritional Services and the Effect on Maternal Weight in an Obese Urban Population
Brief Title: Access to Nutritional Services and the Effect on Maternal Weight Gain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Abington Memorial Hospital (Other)
Responsible Party: Principal Investigator, Erin M. Murphy, MD, Principal Investigator, Abington Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 11-070
Record Dates: First submitted 2012-09-06; First posted 2012-10-25 (Estimated); Last update posted 2013-04-22 (Estimated); Status verified 2013-04

CONDITIONS: Pregnancy; Obesity
Keywords: Pregnancy; Obesity; Nutrition therapy
MeSH Terms: conditions — Obesity | interventions — Nutrition Assessment

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Routine Obstetric Care (No Intervention)
- Nutritional Counseling (Experimental): Patients will receive an initial 90 minute nutritional consult followed by 60 minute follow up consults every 2 weeks to monitor weight gain and nutritional status.
  Interventions: Behavioral: Nutritional Counseling

INTERVENTIONS:
Behavioral: Nutritional Counseling — Patients will keep a daily diary of nutritional intake as well as physical activity. They will also follow up with the nutritional counselor six weeks postpartum.
  Arms: Nutritional Counseling

SUMMARY:
The purpose of this study is to evaluate the effect of access to nutrition services on pregnancy outcomes in the obese urban population. There are many studies that have shown that obesity has a negative impact on pregnancy. However, currently there are only a few small studies that specifically look at ease of access to nutrition services in an obese urban population and the effect this has on maternal weight gain and pregnancy outcomes. This study will compare two groups of pregnant women with a BMI of 30 or greater. The investigators hypothesize that access to nutritional services will lead to decreased weight gain during pregnancy and improved pregnancy outcomes.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the effect of access to nutrition services on pregnancy outcomes in the obese urban population. Approximately one fourth of women in the United States are overweight and nearly one third are considered to be obese. Pregnancy places obese women at increased risk for several adverse events in the antepartum, intrapartum, and postpartum period. There are many studies that have shown that obesity in pregnancy has a negative impact on pregnancy. However, currently there are few studies in the United States that specifically look at ease of access to nutrition services in an obese urban population and the effect this has on pregnancy outcomes. This study will be a randomized controlled study that will compare two groups of pregnant women with a BMI of 30 or greater one of which has access to nutritional services along with routine prenatal care while the other gets only routine prenatal care. The investigators hypothesize that the obese parturient who has access to nutritional services will have decreased weight gain during pregnancy and ultimately have improved pregnancy outcomes. This will help to guide future care for the obese parturient in the urban population who may have limited access to services.

ELIGIBILITY:
Inclusion Criteria:

* primigravid women
* age 19-40yrs
* less than or equal to 18 weeks gestation at time of enrollment
* body mass index (BMI) greater than or equal to 30

Exclusion Criteria:

* multiparous women
* less than 19 yrs of age or older than 40
* greater than 18 weeks gestation at time of enrollment
* body mass index (BMI) less than 30
* any significant past medical history including hypertension, diabetes, renal disease, coagulopathy
* past surgical history of gastric bypass/weight loss surgery

Ages: 19 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2012-12; Primary Completion 2013-12 (Estimated); Study Completion 2014-02 (Estimated)

PRIMARY OUTCOMES:
Weight gain | one year
  change in weight from baseline prepregnancy weight

SECONDARY OUTCOMES:
Birth weight | 40 weeks
  Weight of infant at the time of birth
Fetal anomalies | 40 weeks
  Ultrasound findings of fetal anomalies or those detected at birth
Hypertensive disease of pregnancy | 40 weeks
  Development of hypertensive disease during pregnancy
Gestational diabetes | 40 weeks
  Development of gestational diabetes
Neonatal intensive care admission | 28 days
  Admission to neonatal intensive care unit
APGAR scores | At birth
  Measurement at birth
Mode of delivery | 40 weeks
  vaginal delivery or cesarean section
Intrauterine Fetal Demise | 40 weeks
  Death of fetus prior to delivery
Neonatal Death | 28 days
  Death of neonate from birth to 28 days of life

CONTACTS AND LOCATIONS:
Overall Officials: Erin M Murphy, MD, Principal Investigator — Abington Memorial Hospital; Bethany Perry, MD, Study Director — Abington Memorial Hospital
Locations (1):
- Abington Memorial Hospital, Abington, Pennsylvania, United States